CLINICAL TRIAL: NCT05287048
Title: A Performance Evaluation Study of Arquer Diagnostics Ltd's MCM5 ELISA (ADXGYNAE) Test to Aid in the Diagnosis of Endometrial Cancer
Brief Title: Evaluation of MCM5 in Postmenopausal Bleeding Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Arquer Diagnostics Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: AQ010
Record Dates: First submitted 2022-03-02; First posted 2022-03-18 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Endometrial Cancer
Keywords: Endometrial cancer; Postmenopausal bleeding; MCM5; Biomarker
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine sediment lysate samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with postmenopausal bleeding: Patients attending a gynaecology clinic for investigation of postmenopausal bleeding and undergoing a transvaginal ultrasound (TVUS).
  Interventions: Diagnostic Test: MCM5 ELISA

INTERVENTIONS:
Diagnostic Test: MCM5 ELISA — ADXGYNAE is a non-invasive ELISA utilising a combination of two monoclonal antibodies for the detection of MCM5 in urine sediment. It is intended to aid in the detection of endometrial cancer in women with postmenopausal bleeding who are suspected of having endometrial cancer. Participants will be asked to provide a urine specimen, which will be centrifuged before the sediment is lysed. The lysed sample will then be tested with the MCM5 ELISA.
  Other Names: ADXGYNAE

SUMMARY:
The objective of this multi-centre, prospective study, is to evaluate the performance of a urine MCM5 ELISA test (ADXGYNAE) in the detection of endometrial cancer in patients with postmenopausal bleeding. Patients attending a gynaecology clinic for investigation of postmenopausal bleeding will be recruited and asked to provide a urine sample to be tested. The results of the MCM5 test will be recorded and compared to the patient's routine investigations to determine the clinical utility of the test as an aid in the diagnosis of endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patients who are at least 1 year post-menopausal i.e. have not had a menstrual period for at least one year
* Patients who, in the opinion of the Investigator, are suitable for standard gynaecological investigations as part of normal clinical practice
* Patients who are, in the opinion of the Investigator, able to understand the purpose of the study and provide a full void urine specimen
* Patients who are able to give voluntary, written informed consent to participate in this study and from whom consent has been obtained

Exclusion Criteria:

* Patients with known symptomatic calculi within the urino-genitary system
* Patients currently undergoing chemotherapy or radiotherapy
* Patients who have previously been diagnosed with bladder or renal cancer who are currently in follow up
* Patients with a medical contraindication to endometrial biopsy
* Patients who do not wish to have an endometrial biopsy even if deemed necessary by the treating physician
* Patients who have had urological instrumentation to the urinary tract within 14 days prior to the test (including catheterisation)
* Patients who have had any gynaecological instrumentation in the previous 14 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with postmenopausal bleeding attending a gynaecology clinic for transvaginal ultrasound, who are suspected of having endometrial cancer.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity and negative predictive value (NPV) of ADXGYNAE will be calculated to establish the diagnostic accuracy for the detection of endometrial cancer. | 1 year
  The MCM5 test result will be compared with data obtained from patient's standard of care clinical investigations, including results from transvaginal ultrasound (TVUS) and endometrial biopsy or hysteroscopy. A definitive diagnosis of endometrial cancer will be confirmed by the presence of histologically proven endometrial cancer on resection/biopsy. Patients who do not have an endometrial biopsy will be followed up at 6 months to identify if further investigations were carried out.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Richard Edmondson, MD, Principal Investigator — Central Manchester NHS Foundation Trust
Locations (1):
- Saint Mary's Hospital, Central Manchester NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stockley J, Akhand R, Kennedy A, Nyberg C, Crosbie EJ, Edmondson RJ. Detection of MCM5 as a novel non-invasive aid for the diagnosis of endometrial and ovarian tumours. BMC Cancer. 2020 Oct 15;20(1):1000. doi: 10.1186/s12885-020-07468-y. PMID 33059604